CLINICAL TRIAL: NCT04403230
Title: Periodontal and Prosthetic Outcomes on Teeth Prepared With Biologically Oriented Preparation Technique: Prospective Clinical Study
Brief Title: Outcomes on Teeth Prepared With BOPT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H1448361523684
Record Dates: First submitted 2020-05-20; First posted 2020-05-27 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2020-05

CONDITIONS: Soft Tissues; Prosthetic; Outcome
Keywords: BOPT; dental preparation; dental crown; zirconia; periodontal health

STUDY DESIGN:
Intervention Model Description: This prospective study included 149 teeth treated using biologically oriented preparation technique (BOPT). The sample (149 teeth) was divided into two groups: Seventy four teeth restored with crowns, and 75 teeth supporting fixed partial dentures (FPD).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical behaviour on teeth prepared without finish line (Experimental): Evaluate the clinical behavior of restorations placed on teeth prepared without finish line, monitoring periodontal status as well as the prostheses to assess stability and treatment predictability.
  Interventions: Procedure: Retreatment of teeth prepared without finish line

INTERVENTIONS:
Procedure: Retreatment of teeth prepared without finish line — Retreatment of teeth treated using biologically oriented preparation technique (BOPT). The sample (149 teeth) was divided into two groups: Seventy four teeth restored with crowns, and 75 teeth supporting fixed partial dentures (FPD).

SUMMARY:
The aim of this study is to evaluate the clinical and biological behavior of full coverage restorations on teeth prepared without finish line in a prospective clinical study.

DETAILED DESCRIPTION:
The purpose is to evaluate the clinical and biological behavior of full coverage restorations on teeth prepared without finish line.

This prospective study included 149 teeth treated using biologically oriented preparation technique (BOPT). The sample (149 teeth) was divided into two groups: Seventy four teeth restored with crowns, and 75 teeth supporting fixed partial dentures (FPD). Restorations were fabricated with zirconium oxide cores and ceramic coverings. Patients attended regular annual check-ups when probe depth, presence of inflammation with bleeding on probing, presence of plaque, gingival thickness, marginal stability, biological or mechanical complications, and the patient's level of satisfaction were registered.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (aged over 18 years).
* non-smokers.
* periodontally healthy or periodontally managed.
* patients who had undergone restoration with fixed prostheses (one-piece crowns or fixed partial dentures FPDs) in the aesthetic zone (incisors, canines, premolars, first molars), which needed to be replaced due to biological, esthetic or some other type of problem.

Exclusion Criteria:

* patients who were smokers.
* patients who presented unmanaged parafunctional habits.
* patients with severe systemic diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-01-01 (Actual); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
A possible periodontal complications | Through study completion, an average of 15 years.
  Analyze periodontal outcome on teeth prepared with biologically oriented preparation technique
biological or mechanical prosthetic complications | Through study completion, an average of 15 years.
  Analyze prosthetic outcome on teeth prepared with biologically oriented preparation technique

SECONDARY OUTCOMES:
Patient's level of satisfaction with treatment assessed by means of a visual analogue scale (VAS). | Through study completion, an average of 15 years.
  Patient's satisfaction was assesed using a ''Visual Analogue Scale'' (VAS). In wich 0 is the the minimum and 10 de maximum value, and whether higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Blanca Serra Pastor, Professor, Principal Investigator — University of Valencia